CLINICAL TRIAL: NCT02589496
Title: Phase II Study of Pembrolizumab in Subjects With Advanced Gastric or Gastroesophageal Junction Adenocarcinoma Who Progressed After First-Line Therapy With Platinum and Fluoropyrimidine: Integration of Molecular Subtypes Through Integrative Genomic Analysis
Brief Title: Study of Pembrolizumab in Subjects With Advanced Gastric or Gastroesophageal Junction Adenocarcinoma Who Progressed After First-Line Therapy With Platinum and Fluoropyrimidine: Integration of Molecular Subtypes Through Integrative Genomic Analysis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jeeyun Lee, MD,PhD,Division of hematology-oncology,Department of medicine, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-09-053
Record Dates: First submitted 2015-10-27; First posted 2015-10-28 (Estimated); Results first posted 2023-05-09 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2022-07

CONDITIONS: Gastric Adenocarcinoma; Gastroesophageal Junction Adenocarcinoma
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- pembrolizumab (Experimental): Cohort A :gastric cancer patients Cohort B : MSI-H gastric cancer patients All Chort receive the following treatment.
  * Pembrolizumab 200 mg every 3 weeks
  Interventions: Drug: pembrolizumab

INTERVENTIONS:
Drug: pembrolizumab — 200 mg every 3 weeks
  Other Names: MK-3475; Keytruda

SUMMARY:
This is a single-arm, single-center, open-label trial of pembrolizumab (MK-3475) in subjects with advanced gastric or gastroesophageal junction (GEJ) adenocarcinoma who have progressed after failure of any combination chemotherapy containing a platinum and a fluoropyrimidine agent.

Approximately 60 subjects will be enrollment to evaluate the efficacy and safety of pembrolizumab.

Enrollment will begin with all subjects without regard for PD-L1 expression status. An evaluable specimen for PD-L1 status must be available and confirmed prior to enrollment.

All study subjects will be evaluated every 6 weeks (+/- 7 days) following the date of IP drug adminstration for the first six months and every 12 weeks (+/- 7 days) thereafter until progression of disease is documented with radiologic imaging (computed tomography or magnetic resonance imaging).

In the expansion cohort (cohort B), it was expanded on the original cohort based on response analysis and will be opened separately.

Of the 5 MSI-high patients who were enrolled on to original cohort, all 5 MSI high GC patients (100% response rate) demonstrated dramatic response rate.

Based on this finding, in order to proven Pembrolizumab's efficacy to specific MSI-H GC population, we would like enroll 20 more patients in cohort B. Based on our screening protocol, the prevalence of MSI-high in GC is about 15 %. Only MSI-high GC patients will be included. All the eligibility will be the same.

DETAILED DESCRIPTION:
Each subject will participate in the trial from the time the subject signs the Informed Consent Form (ICF) through the final contact. After a screening phase of up to 28 days, eligible subjects will receive treatment beginning on Day 1 of each 3-week dosing cycle for pembrolizumab.

Treatment with pembrolizumab or paclitaxel will continue until documented disease progression, unacceptable adverse event(s), undercurrent illness that prevents further administration of treatment, Investigator's decision to withdraw the subject, subject withdraw consent, pregnancy of the subject, noncompliance with trial treatment o procedure requirements, subject receives 24 months of pembrolizumab, or administrative reasons requiring cessation of treatment. After the end of treatment, each subject will be followed for 30 days for adverse event monitoring (serious adverse events and events of clinical interest will be collected for 90 days after the end of treatment or 30 days after the end of treatment if the subject initiates new anticancer therapy, whichever is earlier).

Subjects within the pembrolizumab arm who discontinue after 24 months of therapy for reasons other than disease progression or intolerability or who discontinue after attaining a CR may be eligible for up to one year of retreatment after they have experienced radiographic disease progression.

Subjects who discontinue for reasons other than disease progression will have post-treatment follow-up for disease status until disease progression, initiating a non-study cancer treatment, withdrawing consent, or becoming lost to follow-up.

All subjects will be followed by telephone for overall survival until death, withdrawal of consent, or the end of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent/assent for the trial. The subject may also provide consent for Biomedical Research. However, the subject may participate in the main trial without participating in Biomedical Research.
2. Be 19 years of age on day of signing informed consent
3. Have histologically or cytologically-confirmed diagnosis of gastric or Gastroesophageal Junction Adenocarcinoma
4. Have metastatic disease or locally advanced, unresectable disease.
5. Has experienced documented objective radiographic or clinical disease progression during or after first-line therapy containing any platinum,fluoropyrimidine doublet.
6. Have measurable disease based on RECIST as determined by investigator. Tumor lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
7. Be willing to provide fresh tissue for biomarker analysis, and, based on the adequacy of the tissue sample quality for assessment of biomarker status. Repeat samples may be required if adequate tissue is not provided. Newly obtained endoscopic biopsy specimens are preferred to archived samples and formalin-fixed, paraffin-embedded block specimens are preferred to slides.
8. Have a performance status of 0 or 1 on the ECOG Performance Scale.
9. Demonstrate adequate organ function, all screening labs should be performed within 10 days of treatment initiation.
10. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
11. Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
12. Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.
13. (Only Cohort B) confirmed as MSI-H via the PCR or IHC staining by institutional standard.

Exclusion Criteria:

1. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
2. Has squamous cell or undifferentiated gastric cancer.
3. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
4. Has a known history of active Bacillus Tuberculosis
5. Hypersensitivity to pembrolizumab or any of its excipients.
6. Has had a prior anti-cancer monoclonal antibody within 4 weeks prior to study Day 1 or who has not recovered from adverse events due to agents administered more than 4 weeks earlier.
7. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered from adverse events due to a previously administered agent.
8. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
9. Has known active central nervous system metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
10. Has active autoimmune disease that has required systemic treatment in the past 2 years. Replacement therapy is not considered a form of systemic treatment.
11. Has known history of, or any evidence of active, non-infectious pneumonitis.
12. Has an active infection requiring systemic therapy.
13. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
14. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
15. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
16. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
17. Has a known history of Human Immunodeficiency Virus
18. Has known active Hepatitis B or Hepatitis C
19. Has received a live vaccine within 30 days of planned start of study therapy.
20. Is or has an immediate family member who is investigational site or staff directly involved with this trial, unless prospective IRB approval (by chair or designee) is given allowing exception to this criterion for a specific subject.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-03-26 (Actual); Primary Completion 2021-12 (Actual); Study Completion 2021-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, Korea, South Korea

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR

RESULTS

PARTICIPANT FLOW:
Groups:
- Pembrolizumab: Cohort A :gastric cancer patients Cohort B : MSI-H gastric cancer patients All Chort receive the following treatment.
  * Pembrolizumab 200 mg every 3 weeks
  pembrolizumab: 200 mg every 3 weeks
Period: Overall Study
Arm/Group | Pembrolizumab
Started | 80
Completed | 80
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 61
Age, Continuous [Median (Full Range); unit: years] | 57 [26 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 61
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 61
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  South Korea | 61
gastric cancer [Count of Participants; unit: Participants] | 61

OUTCOME MEASURES:

1. Primary Outcome: RR
Description: Objective: To evaluate RR per mRECIST in advanced gastric or GEJ adenocarcinoma who have progressed on one previous line of therapy, when treated with pembrolizumab Hypothesis: Pembrolizumab increases RR per mRECIST with advanced gastric or GEJ adenocarcinoma who have progressed on 1 previous line of therapy
Time Frame: up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 61
Participants | 15

2. Primary Outcome: Response Rate
Description: response rate per RECIST 1.1
Time Frame: 2 years
Population: metastatic gastric cancer patients who failed to standard cytototic chemotherapy
Measure: Count of Participants; unit: Participants
Groups:
- Pembrolizumab: Cohort A :gastric cancer patients
  All Chort receive the following treatment.
  * Pembrolizumab 200 mg every 3 weeks
  pembrolizumab: 200 mg every 3 weeks
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 61
Participants | 15

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 25/61
Serious Adverse Events (participants affected / at risk) | 0/61
Other Adverse Events (participants affected / at risk) | 25/61
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab (N=61)
rash (Skin and subcutaneous tissue disorders) | 2 (2)
pruritis (Skin and subcutaneous tissue disorders) | 7 (7)
nausea (Gastrointestinal disorders) | 4 (4)
diarrhea (Gastrointestinal disorders) | 2 (2)
peripheral sensory neuropathy (Nervous system disorders) | 5 (5)
myalgia (General disorders) | 1 (1)
elevated liver enzyme (Hepatobiliary disorders) | 2 (2)
arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
dry mouth (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-09-10): https://cdn.clinicaltrials.gov/large-docs/96/NCT02589496/Prot_SAP_000.pdf